CLINICAL TRIAL: NCT06510686
Title: Comparison of the Effects of Core Stabilization and Inspiratory Muscle Training on Diaphragm Activation, Inspiratory Muscle Strength, Functional Capacity, Respiratory Functions, Physical Activity and Quality of Life in Patients With COPD
Brief Title: Effects of Core Stabilization and Inspiratory Muscle Training in Patients With COPD
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Ertuğrul Yaşa (Other)
Responsible Party: Sponsor-Investigator, Mustafa Ertuğrul Yaşa, assistant professor, Gulhane School of Medicine
Organization: Gulhane School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-183
Record Dates: First submitted 2024-07-03; First posted 2024-07-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İnspiratory muscle training (Other): Inspiratory muscle training during 8 weeks
  Interventions: Other: İnspiratory muscle training
- Core Stabilization (Other): Inspiratory muscle training and core training during 8 weeks
  Interventions: Other: İnspiratory muscle training; Other: Core training

INTERVENTIONS:
Other: İnspiratory muscle training — exercises to strengthen inspiratory muscles
  Other Names: Normal breath exercises and İnspiratory muscle training
Other: Core training — exercises to strengthen inspiratory and core muscles
  Other Names: Normal breath exercises and İnspiratory muscle training and Core Stabilization
  Arms: Core Stabilization

SUMMARY:
In Chronic Obstructive Pulmonary Disease (COPD), a mismatch develops between the respiratory system's demand and the functional capacity of respiratory muscles due to the combination of local and systemic factors increasing the respiratory workload. This results in impaired coordination of muscle groups, leading to muscle dysfunction. Respiratory muscle dysfunction is a significant determinant of life expectancy in COPD. Additionally, respiratory muscles unable to cope with increased workloads lead to impaired respiratory functions and reduced exercise capacity.

It is widely accepted that appropriate training of respiratory muscles can increase their strength, endurance, and their close relationship with lung volume capacities. Besides their role in respiration, respiratory muscles also contribute to postural function and core stabilization. Studies on respiratory muscle training in COPD have primarily focused on inspiratory muscle strength training, neglecting the core stabilization function of respiratory muscles. However, optimal gains in a muscle can only be achieved with training tailored to its functional characteristics. Therefore, a comprehensive training program should be developed considering the multifunctional nature of respiratory muscles. Studies published in healthy individuals and different patient populations demonstrate that core training can improve lung functions. The aim of this study is to compare the effects of inspiratory muscle training and core stabilization training on diaphragm activation, inspiratory muscle strength, functional capacity, respiratory functions, physical activity, and quality of life in individuals with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Having a diagnosis of COPD according to the GOLD criteria and being at stage 3 or lower
* Not being in an acute exacerbation period and having at least one month since the last exacerbation
* Being able to walk independently
* Having sufficient mental capacity to understand the tasks in the study (Mini-Mental Test >24)
* Being willing to participate in the study

Exclusion Criteria:

* Being a stage 4 COPD patient according to the GOLD criteria
* Having a diagnosis of lung cancer, pulmonary hypertension, and heart failure
* Being in a COPD exacerbation period
* Scoring below 24 on the Mini-Mental Test
* Having any other disease that affects respiratory functions
* Having undergone pulmonary surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-03 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Inspiratory Muscle Strength | 8 weeks
  Maximal Inspiratory Pressure (MIP) (cmH2O),
Inspiratory Muscle Activation | 8 weeks
  surface EMG (TLC from FRC (TLC maneuver)(cmH2O)
Respiratory function tests FEV1 | 8 weeks
  Spirometry, FEV1 (lt)
Respiratory function tests FVC | 8 weeks
  Spirometry, FVC (lt)
Respiratory function tests PEF | 8 weeks
  Spirometry, PEF (lt/sn)
Respiratory function tests FEV1/FVC | 8 weeks
  Spirometry, FEV1/FVC %
Respiratory function MVV | 8 weeks
  Spirometry, MVV(L/min)
Functional capacity | 8 weeks
  Six Minute Walking Test (6MVT) (m)
Symptoms | 8 weeks
  MMRC Dyspnea Scale (Scores range from 0 to 4)

SECONDARY OUTCOMES:
Physical activity, | 8 week
  IPAQ (MET/minute)
Quality of life Tests | 8 week
  SGRQ (Scores range from 0 to 100)
Core Strength | 8 week
  1 minute sit to stand ( how many times sit and stand during 1 minute)
Core Strength flexion | 8 week
  Mcgill Endurance Tests For Trunk Flexion (sec)
Core Strength extension | 8 week
  Mcgill Endurance Tests For Trunk Extension (sec)
Core Strength side bridge | 8 week
  Mcgill Endurance Tests For Side Bridge (sec)

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi, Ankara, Turkey (Türkiye)